CLINICAL TRIAL: NCT03627078
Title: The Effect of Motor Interference Therapy In Traumatic Memories: A Controlled Clinical Trial
Brief Title: Motor Interference Therapy For Traumatic Memories
Acronym: TIMCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez (Other)
Responsible Party: Principal Investigator, Edgar Daniel Crail Melendez, M.SC., El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69/17
Record Dates: First submitted 2018-08-08; First posted 2018-08-13 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Trauma, Psychological; Post Traumatic Stress Disorder
Keywords: traumatic memories; post traumatic stress disorder; motor interference therapy; non pharmacological therapy; trauma related disorders
MeSH Terms: conditions — Psychological Trauma; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Interference Therapy (Experimental): Initial interview applying the Spanish version of the PTSD Symptom Severity Scale-Revised (EGS-R), the visual analogue scale (EQ-VAS) from EuroQol 5D (EQ-5D), and a simple visual-analogue scale (VAS). After that, patients will listen to an audio track twice and follow the instructions. The first four minutes of the audio track instruct the subjects to tap their fingers in response to specific sounds. During the remaining ten minutes, the patients will be asked to recall a traumatic memory while simultaneously are tapping their fingers. Patients must complete at least 80% of the motor task in order to be included. We will reassess a week, a month and six months after the intervention, using all three scales.
  Interventions: Other: motor interference therapy
- Relaxation Exercise (Sham Comparator): Initial interview applying the Spanish version of the PTSD Symptom Severity Scale-Revised (EGS-R), the visual analogue scale (EQ-VAS) from EuroQol 5D (EQ-5D), and a simple visual-analogue scale (VAS). After that, patients will listen to an audio track twice and follow the instructions. The first four minutes of the audio track instruct the subjects in how to do the exercises. During the remaining 10 minutes will hear commands for performing progressive muscle tension-relaxation exercises while the patient evoked the traumatic memory. Patients must complete at least 80% of the motor task in order to be included. We will reassess a week, a month and six months after the intervention, using all three scales.
  Interventions: Other: Relaxation exercises

INTERVENTIONS:
Other: motor interference therapy
  Other Names: TIM
  Arms: Motor Interference Therapy
Other: Relaxation exercises — In a top-down sequence, beginning with the upper body and proceeding to the lower parts. patients contract and relax a specific muscle group following the instructions given by the audio track. We use a shorter version that excludes the legs because of the time.
  Other Names: Jacobson´s progressive relaxation
  Arms: Relaxation Exercise

SUMMARY:
The aim of the study is to compare the effect of motor interference therapy (TIM) to reduce the intensity of discomfort (distress) generated by a traumatic memory compared to a relaxation control maneuver, immediately after the intervention, a week, a month and six months after intervention.

DETAILED DESCRIPTION:
The investigators treated 10 patients with autobiographical traumatic memories using finger tapping tasks, (Motor Interference Therapy <TIM>)in a pilot study with amazing results and a solid size effect. The investigators decided to challenge the intervention using a control task (Jacobson´s progressive relaxation exercises) The hypothesis consists in achieving a 30% reduction of the distress, (measured with Visual Analogue Scale) by using TIM compared with the control task. Patients with traumatic memories will be enrolled in to one of two treatment modalities. The first group will receIve motor interference therapy and the second group will receive a control task (relaxation exercises). Both groups will be assessed using the Spanish version of the PTSD Symptom Severity Scale-Revised (EGS-R), the visual analogue scale (EQ-VAS) from EuroQol 5D (EQ-5D), and a simple visual-analogue scale (VAS) immediately after, a week after, a month after and six months after the treatment for follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 16 years
* Spanish as a native language
* Give written informed consent
* having at least 1 traumatic memory causing distress

Exclusion Criteria:

* Neurological or psychiatric disorders that affect the capacity of verbal comprehension and judgment, such as dementia, psychosis, mental retardation or other cognitive alteration that does not allow them to perform the tasks indicated in the TIM or SHAM
* History of recent substance abuse
* Patients with significant hearing loss or some other hearing impairment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale (EVA) | baseline, immediately, 1 week, 1 month, 6 months
  measures the distress related to traumatic memories in 1-10

SECONDARY OUTCOMES:
Spanish version of the PTSD Symptom Severity Scale-Revised (EGS-R) | baseline, 1 week, 1 month, 6 months
  Posttraumatic stress disorder scale
visual analogue scale (EQ-VAS) from EuroQol 5D (EQ-5D) | baseline, 1 week, 1 month, 6 months
  as a gauge of health-related quality of lif

CONTACTS AND LOCATIONS:
Overall Officials: Edgar D Crail-Melendez, MD, Principal Investigator — El Instituto Nacional de Neurologia y Neurocirugia Manuel Velasco Suarez
Locations (1):
- Instituto Nacional de Neurologia Y Neurocirugia Mvs, Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Morales-Rivero A, Crail-Melendez D, Reyes-Santos L, Bisanz E, Bisanz J, Ruiz-Chow A, Chavarria-Medina MM. Effect of Motor Interference Therapy on Distress Related to Traumatic Memories: A Randomized, Double-Blind, Controlled Feasibility Trial. Brain Behav. 2024 Sep;14(9):e70063. doi: 10.1002/brb3.70063. PMID 39317994